CLINICAL TRIAL: NCT06097702
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BX-001N After Intravenous Administration in Healthy Participants
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of BX-001N in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bilix Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BX-001N-001
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Ischemia-reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BX-001N Part 1 (Experimental): Part 1 is SAD with 5 cohorts where each participant will receive single IV bolus following a 8hr fast.
  Interventions: Drug: BX-001N Part 1
- BX-001N Part 2 (Experimental): Part 2 is MAD with 3 cohorts where each participant will receive 4 sequential daily IV bolus doses following a 8hr fast.
  Interventions: Drug: BX-001N Part 2
- Placebo (Placebo Comparator): Matching doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BX-001N Part 1 — Dosage form- IV bolus Dosage- In the five cohorts, each participant receives a single IV bolus administration in one of the five doses based on body weight and followed up for 7 days.
  Arms: BX-001N Part 1
Drug: BX-001N Part 2 — Dosage form- IV bolus Dosage- In the three cohorts, each participant receives a single IV bolus administration for 4 sequential days in one of the three doses based on body weight and followed up for 14 days.
  Arms: BX-001N Part 2
Drug: Placebo — Participants will receive matching placebo across Part 1 and 2 of the study.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single and multiple ascending dose, Phase 1 study to evaluate the safety, tolerability, and pharmacokinetics of BX-001N after intravenous administration in approximately 64 healthy participants

DETAILED DESCRIPTION:
This study comprises of 2 parts:

* Part 1- Single Ascending Dose (SAD)- This part will enroll approximately 40 participants across 5 cohorts where each participant will receive a single intravenous (IV) bolus dose in healthy participants. On Day 1, participants in each cohort will receive investigational product (IP) (i.e., BX-001N or Placebo) as a single IV bolus following a minimum 8-hour fast.
* Part 2 -Multiple Ascending Dose (MAD)- This part will enroll approximately 24 participants across 3 cohorts where each participants will receive intravenous (IV) bolus dose for 4 sequential daily. At the same time each morning from Day 1 to Day 4 (inclusive), participants in each cohort will receive IP (i.e., BX-001N or Placebo) as a single IV bolus following a minimum 8-hour fast.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age
* In good general health at Screening and/or before the first administration of IP
* BMI > 18.0 and < 32.0 kg/m2 at Screening
* Nonsmoker and must not have used any tobacco products within 2 months prior to screening
* Females must not be pregnant or lactating, and females and males must use acceptable, highly effective double contraception during study and follow-up period
* Person who can provide written informed consent prior to the commencement of all study procedures

Exclusion Criteria:

* Underlying physical or psychological medical condition to comply with the protocol or complete the study per protocol
* Genetic disorder with severe and abnormal bilirubin metabolism
* Blood or plasma donation or significant blood loss prior to the first administration of IP
* Viral or bacterial infection prior to the first administration of IP
* Poor venous access
* Significant scarring or tattoos at the planned site of IP administration
* History of severe allergic or anaphylactic reactions, or sensitivity to the IP or its constituents
* History or active cardiovascular, respiratory, kidney, endocrine, blood, digestive, central nervous, urinary and/or musculoskeletal disease
* History of malignancy prior to Screening
* Abnormal ECG findings
* History or presence of a condition associated with significant immunosuppression
* History of life-threatening infection
* Infections requiring parenteral antibiotics
* Vaccination prior to the first administration of IP
* Exposure to any significantly immune suppressing drug
* Abnormal vital signs findings
* Abnormal laboratory findings
* Positive results for viral testing at Screening
* Positive result at Screening and Day -1 for toxicology screening panel
* History of substance abuse or dependency or history of recreational intravenous (IV) drug use
* Excess of regular alcohol consumption
* Use of any IP or investigational medical device within 30 days prior to Screening
* Unable to adhere to the prohibited therapies
* Unwilling to adhere to the dietary restrictions
* Unwilling to refrain from strenuous exercise

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment emergent Adverse events (TEAEs) | SAD-Screening to Day 7; MAD- Screening to Day 14
  TEAE will be collected to assess participants' safety after BX-001N treatment
Number of participants with clinical laboratory abnormalities | SAD-Screening to Day 7; MAD- Screening to Day 14
Number of participants with changes in the 12-lead electrocardiogram (ECG) | SAD-Screening to Day 7; MAD- Screening to Day 14
Number of incidences of injection site reactions | SAD-Day 1 to Day 2; MAD- Day 1 to Day 5

SECONDARY OUTCOMES:
Changes in Cmax (maximum Concentration) of BX-001N with 5 different doses of SAD and 3 different doses of MAD | SAD- Day 1 to Day 7; MAD- Day 1 to Day 14
  SAD's samples of PK are collected at total 14 time points up to Day 7 post dose. MAD's samples of PK are collected at total 26 time points from pre-dose and up to day 14 after dosing.
Changes in Tmax (Time of maximum Concentration) of BX-001N with 5 different doses of SAD and 3 different doses of MAD | SAD- Day 1 to Day 7; MAD- Day 1 to Day 14
  SAD's samples of PK are collected at total 14 time points up to Day 7 post dose. MAD's samples of PK are collected at total 26 time points from pre-dose and up to day 14 after dosing.
Changes in AUC (area under curve) of BX-001N with 5 different doses of SAD and 3 different doses of MAD | SAD- Day 1 to Day 7; MAD- Day 1 to Day 14
  SAD's samples of PK are collected at total 14 time points up to Day 7 post dose. MAD's samples of PK are collected at total 26 time points from pre-dose and up to Day 14 after dosing.
Change in Immunogenicity- Incidence of Anti-drug antibody (ADA) by polyethylene glycol (PEG) | SAD-Day 1 to Day 7; MAD- Day 1 to Day 14
  Up to 3 samples will be collected in total and additional samples if positive results
Change in Immunogenicity- Titers of Anti-drug antibody (ADA) by polyethylene glycol (PEG) | SAD-Day 1 to Day 7; MAD- Day 1 to Day 14
  Up to 3 samples will be collected in total and additional samples if positive results
Change in Immunogenicity- Duration of Anti-drug antibody (ADA) by polyethylene glycol (PEG) | SAD-Day 1 to Day 7; MAD- Day 1 to Day 14
  Up to 3 samples will be collected in total and additional samples if positive results

CONTACTS AND LOCATIONS:
Overall Officials: Angela C Rowland, Dr, Principal Investigator — CMAX Clinical Research
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No